CLINICAL TRIAL: NCT06084481
Title: A Phase 1 Open-Label Study to Evaluate the Efficacy and Safety of ABBV-400 in Select Advanced Solid Tumor Indications
Brief Title: Study to Assess Adverse Events and Change in Disease Activity in Adult Participants With Select Advanced Solid Tumor Indications Receiving Intravenous (IV) ABBV-400
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M24-427; 2023-506227-29-00 (Other: EU CT)
Record Dates: First submitted 2023-10-10; First posted 2023-10-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Hepatocellular Carcinoma; Pancreatic Ductal Adenocarcinoma; Biliary Tract Cancers; Esophageal Squamous Cell Carcinoma; Triple Negative Breast Cancer; Hormone Receptor+/Human Epidermal Growth Factor Receptor 2 Negative Breast Cancer; Head and Neck Squamous-Cell Carcinoma; Platinum Resistant High Grade Epithelial Ovarian Cancer
Keywords: Hepatocellular Carcinoma; Pancreatic Ductal Adenocarcinoma; Biliary Tract Cancers; Esophageal Squamous Cell Carcinoma; Triple Negative Breast Cancer; Hormone Receptor+/Human Epidermal Growth Factor Receptor 2 Negative Breast Cancer; Head and Neck Squamous-Cell Carcinoma; Platinum Resistant High Grade Epithelial Ovarian Cancer; Solid Tumors; Advanced Solid Tumors; ABBV-400
MeSH Terms: conditions — Carcinoma, Hepatocellular; Biliary Tract Neoplasms; Esophageal Squamous Cell Carcinoma; Triple Negative Breast Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- Cohort 1: Hepatocellular Carcinoma (HCC) (Experimental): Participants with HCC will receive ABBV-400 for up to 3 years during and up to the treatment period with an additional safety follow-up period of up to 2 years.
  Interventions: Drug: ABBV-400
- Cohort 2: Pancreatic Ductal Adenocarcinoma (PDAC) (Experimental): Participants with PDAC will receive ABBV-400 for up to 3 years during and up to the treatment period with an additional safety follow-up period of up to 2 years.
  Interventions: Drug: ABBV-400
- Cohort 3: Biliary Tract Cancers (BTC) (Experimental): Participants with BTC will receive ABBV-400 for up to 3 years during and up to the treatment period with an additional safety follow-up period of up to 2 years.
  Interventions: Drug: ABBV-400
- Cohort 4: Esophageal Squamous Cell Carcinoma, (ESCC) (Experimental): Participants with ESCC will receive ABBV-400 for up to 3 years during and up to the treatment period with an additional safety follow-up period of up to 2 years.
  Interventions: Drug: ABBV-400
- Cohort 5: Triple Negative Breast Cancer (TNBC) (Experimental): Participants with TNBC will receive ABBV-400 for up to 3 years during and up to the treatment period with an additional safety follow-up period of up to 2 years.
  Interventions: Drug: ABBV-400
- Cohort 6: Hormone Receptor+/HER2-breast Cancer (HR+/HER2-BC) (Experimental): Participants with HR+/HER2-BC will receive ABBV-400 for up to 3 years during and up to the treatment period with an additional safety follow-up period of up to 2 years.
  Interventions: Drug: ABBV-400
- Cohort 7: Head and Neck Squamous-cell-carcinoma (HNSCC) (Experimental): Participants with HNSCC will receive ABBV-400 for up to 3 years during and up to the treatment period with an additional safety follow-up period of up to 2 years.
  Interventions: Drug: ABBV-400
- Cohort 8: PROC/Primary Peritoneal/Fallopian Tube Cancer (Experimental): Participants with Platinum Resistant High Grade Epithelial Ovarian Cancer (PROC)/primary peritoneal/fallopian tube cancer will receive ABBV-400 for up to 3 years during and up to the treatment period with an additional safety follow-up period of up to 2 years.
  Interventions: Drug: ABBV-400
- Cohort 9: Drug-Drug Interaction (Experimental): Participants with advanced or metastatic solid tumors will receive ABBV-400 and a strong CYP3A4 inhibitor (ITZ) for up to 3 years during and up to the treatment period with an additional safety follow-up period of up to 2 years.
  Interventions: Drug: ABBV-400; Drug: Itraconazole (ITZ)

INTERVENTIONS:
Drug: ABBV-400 — Intravenous (IV) Infusion
Drug: Itraconazole (ITZ) — Oral Solution
  Arms: Cohort 9: Drug-Drug Interaction

SUMMARY:
Cancer is a condition where cells in a specific part of body grow and reproduce uncontrollably. The purpose of this study is to assess adverse events and change in disease activity when ABBV-400 is given to adult participants to treat advanced solid tumors.

ABBV-400 is an investigational drug being developed for the treatment of advanced solid tumors. Study doctors put the participants in groups called cohorts. Cohorts 1-8 receive ABBV-400 alone (monotherapy) followed by a safety follow-up period. Cohort 9 receives ABBV-400 in combination with a strong CYP3A3 inhibitor (ITZ) followed by a safety follow-up period. Approximately 285 adult participants with hepatocellular carcinoma (HCC), pancreatic ductal adenocarcinoma (PDAC), biliary tract cancers (BTC), esophageal squamous cell carcinoma (ESCC), triple negative breast cancer (TNBC), hormone receptor+/human epidermal growth factor receptor 2 negative (HER2-) breast cancer (hormone receptor-positive [HR+]/HER2-breast cancer [BC]), head and neck squamous-cell-carcinoma (HNSCC), Platinum Resistant High Grade Epithelial Ovarian Cancer (PROC)/primary peritoneal/fallopian tube cancer, or advanced solid tumors, will be enrolled in the study in approximately 54 sites worldwide.

In cohorts 1-8, participants with the following advanced solid tumor indications: HCC, PDAC, BTC, ESCC, TNBC, HR+/HER2-BC, HNSCC, and PROC/primary peritoneal/fallopian tube cancer will receive intravenous (IV) ABBV-400 monotherapy and in cohort 9 participants will receive intravenous (IV) ABBV-400 and an oral solution of ITZ, for up to 3 years during and up to the treatment period with an additional safety follow-up period of up to 2 years.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at an approved institution (hospital or clinic). The effect of the treatment will be frequently checked by medical assessments, blood tests, questionnaires and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory values meeting the criteria laid out in the protocol.
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
* Documented diagnosis of locally advanced or metastatic hepatocellular carcinoma (HCC), pancreatic ductal adenocarcinoma (PDAC), biliary tract cancers (BTC), squamous cell carcinoma of the esophagus, (ESCC), triple negative breast cancer (TNBC), hormone receptor+/HER2-breast cancer (HR+/HER2-BC), head and neck squamous-cell-carcinoma (HNSCC), or Platinum Resistant High Grade Epithelial Ovarian Cancer (PROC)/primary peritoneal/fallopian tube cancer (by World Health Organization [WHO] criteria). Participant meets the criteria for disease activity laid out in the protocol.

Exclusion Criteria:

* Have received anticancer therapy including chemotherapy, radiation therapy, immunotherapy, biologic, or any investigational therapy within 28 days or 5 half-lives of the drug (whichever is shorter) prior to the first dose of ABBV-400. Palliative radiation therapy for bone, skin, or subcutaneous metastases with 10 fractions or less is permitted and not subject to a washout period.
* Unresolved clinically significant AEs > Grade 1 from prior anticancer therapy.
* History of interstitial lung disease (ILD) or pneumonitis that required treatment with systemic steroids, or any evidence of active ILD or pneumonitis, including but not limited to those listed in the protocol.
* History of clinically significant, intercurrent lung-specific illnesses, including those laid out in the protocol.
* Untreated brain or meningeal metastases (i.e., participants with history of metastases are eligible provided they do not require ongoing steroid treatment for cerebral edema and have shown clinical and radiographic stability for at least 14 days after definitive therapy). Participants may continue on antiepileptic therapy if required.
* History of other active malignancy, with the exception of those laid out in the protocol.
* Any autoimmune, connective tissue or inflammatory disorders with documented or suspicious pulmonary involvement at screening (i.e., rheumatoid arthritis, Sjogren's, sarcoidosis etc.), and prior pneumonectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2023-11-09 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 36 Months
  ORR defined as percentage of participants with confirmed best overall response of confirmed partial response (PR) or better per investigator review according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Number of Participants with Adverse Events (AEs) | Up to 36 Months
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation in which a participant is administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.
Maximum Observed Concentration (Cmax) of ABBV-400 Conjugate | Up to 36 Months
  Cmax of ABBV-400 conjugate.
AUC from Time 0 to the End of Dosing Interval (AUCtau) of ABBV-400 Conjugate | Up to 36 Months
  AUCtau of ABBV-400 conjugate.

SECONDARY OUTCOMES:
Duration of Response (DOR) for Participants with Confirmed Complete Response (CR)/PR | Up to 36 Months
  DOR is defined for participants achieving a confirmed PR or better as the time from the initial response of PR (or better) per investigator review according to RECIST 1.1 criteria to disease progression or death of any cause, whichever occurs earlier.
Clinical Benefit Rate | Up to 36 Months
  CBR is defined as the proportion of participants with a best overall response of stable disease at least 5 weeks post first dose, confirmed CR or PR per investigator review according to RECIST, version 1.1
Progression-free Survival (PFS) | Up to 36 Months
  PFS is defined as time from first study treatment to a documented disease progression according to RECIST, version 1.1, as determined by the investigator, or death due to any cause, whichever occurs earlier.
Overall Survival (OS) | Up to 36 Months
  OS is defined as time from first study treatment to death due to any cause.
Cmax of ABBV-400 | Up to 36 Months
  Cmax of ABBV-400.
Time to Cmax (Tmax) of ABBV-400 | Up to 36 Months
  Tmax of ABBV-400.
Area Under the Plasma Concentration-time Curve (AUC) for Total Antibody Concentration | Up to 36 Months
  AUC for total antibody concentration.
Total Antibody Drug Conjugate (ADC) Concentration | Up to 36 Months
  Total ADC concentration.
Plasma Concentrations of Unconjugated Topoisomerase 1 (Top1) Inhibitor Payload | Up to 36 Months
  Plasma concentrations of unconjugated Top1 inhibitor payload.
Antidrug Antibody (ADA) | Up to 36 Months
  Incidence and concentration of anti-drug antibodies.
Neutralizing Antidrug Antibody (nADA) | Up to 36 Months
  Incidence and concentration of neutralizing anti-drug antibodies.
Tmax of ABBV-400 Conjugate | Up to 36 Months
  Tmax of ABBV-400 conjugate.
Tmax of ABBV-400 Unconjugated | Up to 36 Months
  Tmax of ABBV-400 unconjugated.
Terminal Phase Elimination Half-Life (t1/2) of ABBV-400 Conjugate | Up to 36 Months
  t1/2 of ABBV-400 conjugate.
t1/2 of ABBV-400 Unonjugated | Up to 36 Months
  t1/2 of ABBV-400 unconjugated.
Volume of Distribution at Steady State (Vss) of ABBV-400 Conjugate | Up to 36 Months
  Vss of ABBV-400 conjugate.
Vss of ABBV-400 Unconjugated | Up to 36 Months
  Vss of ABBV-400 unconjugated.
Total Body Clearance at Steady State (CLss) of ABBV-400 Conjugate | Up to 36 Months
  CLss of ABBV-400 conjugate.
CLss of ABBV-400 Unconjugated | Up to 36 Months
  CLss of ABBV-400 unconjugated.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (54):
- United States (20):
  - City of Hope National Medical Center /ID# 258645, Duarte, California
  - Ucsf /Id# 257705, San Francisco, California
  - University of Colorado Cancer Center - Cancer Clinical Trials Office /ID# 255128, Aurora, Colorado
  - Sarah Cannon Research Institute at HealthONE - Denver /ID# 258926, Denver, Colorado
  - Florida Cancer Specialists /ID# 261569, Sarasota, Florida
  - Northwestern University Feinberg School of Medicine /ID# 257378, Chicago, Illinois
  - University of Chicago Medical Center /ID# 258197, Chicago, Illinois
  - START Midwest /ID# 256581, Grand Rapids, Michigan
  - Washington University-School of Medicine /ID# 257379, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center-Koch Center /ID# 255132, New York, New York
  - Duke Cancer Center /ID# 255129, Durham, North Carolina
  - Univ Hosp Cleveland /ID# 257706, Cleveland, Ohio
  - Lifespan Cancer Institute at Rhode Island Hospital /ID# 257693, Providence, Rhode Island
  - MUSC Hollings Cancer Center /ID# 257935, Charleston, South Carolina
  - Prisma Health /ID# 257697, Greenville, South Carolina
  - Tennessee Oncology-Nashville Centennial /ID# 261568, Nashville, Tennessee
  - MD Anderson Cancer Center /ID# 255131, Houston, Texas
  - Univ Texas HSC San Antonio /ID# 257708, San Antonio, Texas
  - South Texas Accelerated Research Therapeutics /ID# 260404, San Antonio, Texas
  - Inova Schar Cancer Institute - Fairfax - Innovation Park Drive /ID# 262771, Fairfax, Virginia
- Australia (2):
  - Chris O'Brien Lifehouse /ID# 262765, Camperdown, New South Wales
  - Austin Health /ID# 256635, Heidelberg, Victoria
- Israel (5):
  - The Chaim Sheba Medical Center /ID# 255731, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 258931, Tel Aviv, Tel Aviv
  - Rambam Health Care Campus /ID# 256649, Haifa
  - Hadassah Medical Center-Hebrew University /ID# 256655, Jerusalem
  - Rabin Medical Center. /ID# 256650, Petah Tikva
- Japan (7):
  - NHO Nagoya Medical Center /ID# 261001, Nagoya, Aichi-ken
  - Aichi Cancer Center Hospital /ID# 256679, Nagoya, Aichi-ken
  - National Cancer Center Hospital East /ID# 258934, Kashiwa-shi, Chiba
  - Kyoto University Hospital /ID# 256680, Kyoto, Kyoto
  - Shizuoka Cancer Center /ID# 257789, Sunto-gun, Shizuoka
  - National Cancer Center Hospital /ID# 261136, Chuo-Ku, Tokyo
  - The Cancer Institute Hospital Of JFCR /ID# 257788, Koto-ku, Tokyo
- Pan American Center for Oncology Trials /ID# 262903, Rio Piedras, Puerto Rico
- South Korea (6):
  - Inje University Haeundae Paik Hospital /ID# 260118, Busan, Busan Gwang Yeogsi
  - Gyeongsang National University Hospital /ID# 260408, Jinju, Gyeongsangnam-do
  - Chungbuk National University Hospital /ID# 256698, Cheongju-si, North Chungcheong
  - Seoul National University Hospital /ID# 255730, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 258933, Seoul, Seoul Teugbyeolsi
  - Korea University Guro Hospital /ID# 256700, Seoul, Seoul Teugbyeolsi
- Spain (9):
  - Institut Català d'Oncologia (ICO) - Badalona /ID# 263954, Badalona, Barcelona
  - Hospital Quirón Málaga /ID# 263994, Málaga, Malaga
  - Clinica Universidad de Navarra - Pamplona /ID# 256703, Pamplona, Navarre
  - Hospital HM Nou Delfos /ID# 263953, Barcelona
  - Hospital General Universitario Gregorio Maranon /ID# 262816, Madrid
  - Clinica Universidad de Navarra - Madrid /ID# 264042, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz /ID# 256702, Madrid
  - Hospital Universitario HM Sanchinarro /ID# 256701, Madrid
  - Hospital Universitario Miguel Servet /ID# 256704, Zaragoza
- Taiwan (4):
  - E-DA Cancer Hospital /ID# 258880, Kaohsiung City, Kaohsiung
  - National Taiwan University Hospital /ID# 256713, Taipei City, Taipei
  - China Medical University Hospital /ID# 256712, Taichung
  - Linkou Chang Gung Memorial Hospital /ID# 259420, Taoyuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-427